CLINICAL TRIAL: NCT05601752
Title: A Phase 2, Open-Label, Randomized, Non-Comparative Clinical Trial of ADP-A2M4CD8 Monotherapy and in Combination with Nivolumab in Subjects with Recurrent Ovarian Cancers
Brief Title: ADP-A2M4CD8 Monotherapy and in Combination with Nivolumab in HLA-A2+ Subjects with MAGE-A4 Positive Ovarian Cancer (SURPASS-3)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0055-003/GOG-3084
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous genetically modified ADP-A2M4CD8 cells (Experimental)
  Interventions: Genetic: Autologous genetically modified ADP-A2M4CD8 cells
- Autologous genetically modified ADP-A2M4CD8 cells in combination with Nivolumab (Experimental)
  Interventions: Combination Product: Autologous genetically modified ADP-A2M4CD8 cells in combination with Nivolumab

INTERVENTIONS:
Genetic: Autologous genetically modified ADP-A2M4CD8 cells — Infusion of autologous genetically modified ADP-A2M4CD8 cells on Day 1
  Arms: Autologous genetically modified ADP-A2M4CD8 cells
Combination Product: Autologous genetically modified ADP-A2M4CD8 cells in combination with Nivolumab — Infusion of autologous genetically modified ADP-A2M4CD8 on Day 1 followed by nivolumab 480 mg IV at Week 4 and then every four weeks
  Arms: Autologous genetically modified ADP-A2M4CD8 cells in combination with Nivolumab

SUMMARY:
This is a phase 2, open-label, randomized, non-comparative clinical trial to evaluate the clinical outcome of ADP A2M4CD8 as monotherapy and in combination treatment with nivolumab in human leukocyte antigen (HLA) A2+ subjects with recurrent ovarian cancer positive for MAGE-A4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be assessed for eligibility prior to leukapheresis AND prior to lymphodepleting chemotherapy (unless otherwise noted) and must meet all specified criteria for study participation.

Inclusion Criteria:

1. Subject (or legally authorized representative) has voluntarily agreed to participate by giving written informed consent in accordance with International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidelines and applicable local regulations.
2. Subject (or legally authorized representative) has agreed to abide by all protocol-required procedures including study related assessments and management by the treating institution for the duration of the study, including LTFU.
3. Subject is ≥ 18 and ≤ 75 years of age at the time the Pre Screening informed consent form (ICF) is signed.
4. Subject has histologically confirmed diagnosis of high-grade serous or high-grade endometrioid recurrent ovarian carcinoma, including primary peritoneal and fallopian tube carcinoma.
5. Subject has measurable disease according to RECIST v1.1 prior to lymphodepletion. Measurable disease is not required prior to leukapheresis.
6. Subject has the following disease-specific prior therapy requirements:

   1. The initial therapy must have included at least 3 cycles of a prior platinum and taxane based chemotherapy regimen for primary disease, possibly including intraperitoneal therapy, consolidation, or extended therapy (maintenance/consolidation).
   2. Subjects may receive up to 4 prior regimens of combination or single agent systemic treatment for their disease, which may include investigational therapies unless discussed and agreed upon with the Sponsor or designee. Note: Neo-adjuvant/adjuvant treatment is considered as one line of treatment. Bridging therapy is permitted and is not considered as a line of treatment.
   3. Subjects who have received only 1 line of platinum based therapy must have progressed between 93 and 183 days of completing platinum based therapy as a part of front line treatment of ovarian cancer. Subjects who have progressed within 92 days of completing platinum based therapy in front line treatment are excluded.
   4. Subjects who have received 2 or more lines of platinum based therapy must have progressed during or within 183 days of completing the latest platinum based therapy for treatment of recurrent ovarian cancer. The number of days (platinum-free interval) should be calculated from the date of the last administered dose of platinum therapy to the date of documentation of progression.
   5. Subjects with a known BRCA mutation (germ line or somatic) must have received a poly adenosine diphosphate-ribose polymerase (PARP).
   6. Subjects must have received bevacizumab.
7. Positive for HLA-A*02:01, HLA-A*02:02, HLA-A*02:03, or HLA-A*02:06 allele as determined by Adaptimmune-designated central laboratory testing. HLA-A*02 alleles having the same protein sequence in the peptide binding domains (P group) will also be included. Other HLA-A*02 alleles may be eligible after adjudication with the Sponsor.
8. MAGE-A4 expression, defined as ≥ 30% of tumor cells that are ≥ 2+ by IHC, should be documented at the pre screening period based on either an archival specimen or a fresh biopsy. All samples must have been pathologically reviewed by an Adaptimmune-designated central laboratory confirming expression.
9. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
10. Subject has left ventricular ejection fraction (LVEF) of ≥ 50% or the institutional lower limit of normal range, whichever is lower.
11. Subject is fit for leukapheresis, and adequate venous access can be established for the cell collection.
12. Subjects of childbearing potential must have a negative urine or serum pregnancy test AND must agree to use a highly effective method of contraception starting at the first dose of chemotherapy and continue for at least 12 months or for 4 months after the gene-modified cells are no longer detected in the blood, or 6 months after the last dose of nivolumab, whichever is longer. Subjects of childbearing potential must also agree to refrain from egg donation, storage, or banking during these same time periods.
13. Subjects must have ≥ 90% room air oxygen saturation test at rest at Screening (within 7 days of leukapheresis) and at Baseline.
14. Subject must have adequate organ function as indicated by the laboratory values in the table below.

System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (without granulocyte colony stimulating factor [G-CSF] support) Platelets ≥ 100 × 109/L (without transfusion support within 5 days prior to leukapheresis and lymphodepletion) Hemoglobin (Hb) ≥ 90 g/L (without transfusion support within 5 days prior to leukapheresis and lymphodepletion) Coagulation Prothrombin time or international normalized ratio (INR) ≤ 1.5 × upper limit of normal (ULN), unless receiving therapeutic anticoagulation Partial thromboplastin time ≤ 1.5 × ULN, unless receiving therapeutic anticoagulation Renal Glomerular filtration rate (GFR) or creatinine clearance (CrCl) (estimated or calculated)1 ≥ 50 mL/min /1.73 m2 or ≥ 50 mL/min Hepatic Serum total bilirubin ≤ 1.5 × ULN (unless subject has documented Gilbert's Syndrome with direct bilirubin < 35% of total bilirubin) Exception: Subjects with liver metastasis ≤ 2.5 × ULN Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST) ≤ 2.5 × ULN Albumin ≥ 3 g/dL (Without albumin deficit replacement within 7 days only prior to leukapheresis) Exception: Subjects with liver metastasis ≤ 5.0 × ULN

1 Renal function (GFR or CrCl) will be estimated or measured according to standard practice at the treating institution. Renal function will be reassessed at Baseline using the same methodology.

Note: Laboratory values that are slightly out of the laboratory test parameters, if assessed as not clinically significant by the site study Investigator, may be acceptable after discussion and review by the Sponsor Study Physician. This applies to screening laboratory assessments and baseline laboratory assessments.

Exclusion Criteria:

1. Positive for HLA-A*02:05 in either allele as determined by Adaptimmune-designated central laboratory testing. HLA-A*02 alleles having the same protein sequence as HLA-A*02:05 in the peptide binding domains (P groups) will also be excluded. Other alleles may be exclusionary after adjudication with the Sponsor.
2. Subject has received or plans to receive the following therapy/treatment prior to to leukapheresis or lymphodepleting chemotherapy, unless stopped according to the washout requirements:

   Cytotoxic chemotherapy Required Washout Prior to Leukapheresis 3 weeks Required Washout Prior to Lymphodepletion: 3 weeks

   Small molecules/tyrosine kinase inhibitors (TKIs), such as dabrafenib, trametinib, vemurafenib, and cobimetinib Note: No washout period is required for compounds that do not cause bone marrow suppression/lymphopenia or for epidermal growth factor receptor and alkaline phosphatase/ ROS 1 inhibitors. Required Washout Prior to Leukapheresis 1 week Required Washout Prior to Lymphodepletion: 1 week

   Immune therapy (including monoclonal antibody therapy, checkpoint inhibitors, and biologics) other than anti-PD(L)1 Required Washout Prior to Leukapheresis 2 weeks Required Washout Prior to Lymphodepletion: 2 weeks

   Anti-PD(L)1 Required Washout Prior to Leukapheresis 2 weeks Required Washout Prior to Lymphodepletion: 6 weeks

   Experimental anti-cancer vaccine Required Washout Prior to Leukapheresis: N/A Required Washout Prior to Lymphodepletion: Eight weeks in the absence of tumor response.

   The subject should be excluded if their disease is responding to an experimental vaccine given within 6 months.

   Gene therapy using an integrating vector Subjects who have received a gene therapy using any DNA-integrating vector other than a lentivirus (retrovirus, Adeno-associated Virus (AAV), etc.) are excluded from this study. Use of previous gene therapy using a lentiviral vector is permitted. If transduced T-cells represent < 1% of PBMCs (< 1500 copies of vectors/μg of PBMC DNA) at the time of screening. Eligibility testing must be done by Adaptimmune's designated Contract Research Organization (CRO). Required Washout Prior to Lymphodepletion: N/A

   Corticosteroids or any other immunosuppressive therapy Note: Use of topical or inhaled steroids is not an exclusion. See Section 6.5.1 for exceptions.

   Required Washout Prior to Leukapheresis: 2 weeks Required Washout Prior to Lymphodepletion 2 weeks

   Anti-MAGE-A4 therapy Note: Fresh screening biopsy post-anti-MAGE-A4 therapy must be obtained to confirm MAGE-A4 positivity by IHC. Required Washout Prior to Leukapheresis: 2 weeks Required Washout Prior to Lymphodepletion: 2 weeks

   Investigational treatment Required Washout Prior to Leukapheresis 2 weeks or 5 half-lives, whichever is shorter Required Washout Prior to Lymphodepletion: 2 weeks or 5 half-lives, whichever is shorter.

   Radiation to vital organs (e.g., liver, kidney) Required Washout Prior to Leukapheresis: N/A Required Washout Prior to Lymphodepletion: 4 weeks

   Radiation to the pelvis Required Washout Prior to Leukapheresis: 4 weeks Required Washout Prior to Lymphodepletion: 4 weeks

   Whole brain radiotherapy (WBRT) or brain stereotactic radiosurgery (SRS) Required Washout Prior to Leukapheresis N/A Required Washout Prior to Lymphodepletion: 2 weeks

   Radiotherapy to the target lesions Required Washout Prior to Leukapheresis: N/A Required Washout Prior to Lymphodepletion: 3 months prior to lymphodepleting chemotherapy or a target lesion with progression post radiotherapy (Note: There is no washout period for palliative radiation to non-target organs.)

   PARP inhibitor Required Washout Prior to Leukapheresis: 1 week Required Washout Prior to Lymphodepletion: 1 week

   Antibody drug conjugates (such as mirvetuximab) Required Washout Prior to Leukapheresis: 3 weeks Required Washout Prior to Lymphodepletion: 3 weeks Note: Duration of any other anti-cancer therapies must be discussed and agreed upon with the Sponsor Study Physician
3. Toxicity from previous anti-cancer therapy that has not recovered to Grade ≤ 1 or baseline prior to enrollment (except for nonclinically significant toxicities, e.g., alopecia and vitiligo). Subjects with Grade 2 toxicities that are deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled.
4. Subject has a history of allergic reactions attributed to compounds of similar chemical or biological composition to fludarabine, cyclophosphamide, or other agents used in the study.
5. Subject has an active autoimmune or immune-mediated disease that has not yet been resolved. Subjects with immune-mediated AEs secondary to treatment with immunotherapy that resolve to Grade ≤ 1 off steroids are permitted. Subjects with hypothyroidism, type I diabetes, adrenal insufficiency, or pituitary insufficiency that are stable on replacement therapy are eligible. Subjects with disorders such as asthma, vitiligo, psoriasis, or atopic dermatitis that are well controlled without requiring systemic immunosuppression are also eligible. Other stable immune conditions that do not require prednisone > 20 mg/day (or its equivalent for other corticosteroid agents) may be acceptable with the agreement of the Sponsor.
6. Subject had major surgery within 4 weeks prior to lymphodepletion; subjects should have been fully recovered from any surgical-related toxicities. Surgical-related toxicities that are not clinically significant per Investigator assessment may be acceptable after discussion and agreement with the Study Physician.
7. Leptomeningeal disease, carcinomatous meningitis, or symptomatic central nervous system (CNS) metastases. Subjects with prior history of symptomatic CNS metastases must have received treatment (i.e., SRS, WBRT, or surgery) and be neurologically stable for at least 1 month, not requiring anti-seizure medications, or off steroids for at least 14 days prior to leukapheresis and lymphodepletion. Subjects who have asymptomatic CNS metastases without associated edema, shift, or requirement for steroids or anti-seizure medications are eligible. If such a subject receives SRS or WBRT, a minimum period of 2 weeks needs to lapse between the therapy and lymphodepletion. Prophylactic anti-seizure medication is allowed.
8. Subject has any other prior malignancy that is not considered by the Investigator to be in complete remission. Resectable squamous or basal cell carcinoma of the skin is acceptable. Prior malignancies that have been surgically resected and show no evidence of disease are acceptable.
9. Clinically significant cardiovascular disease including, but not limited to, any of the following:

   1. Electrocardiogram (ECG) showing clinically significant abnormality at Screening
   2. Uncontrolled clinically significant arrhythmias
   3. Known family history or congenital history of prolonged QT syndrome or history of torsade de pointes
   4. Uncontrolled hypertension despite optimal medical therapy
   5. Acute coronary syndrome (angina or myocardial infarction) in the last 6 months
   6. Clinically significant cardiac disease defined by congestive heart failure New York Heart Association Class 3 and 4
   7. History of stroke, CNS bleeding, transient ischemic attack, or reversible ischemic neurologic deficit within last 6 months
10. Uncontrolled intercurrent illness including, but not limited to, any of the following:

    1. Ongoing or active systemic infection, or localized infection which may become systemic due to leukapheresis procedure, e.g., catheter insertion will be excluded. Subjects with urinary tract infections will be included only following treatment with antibiotics.(For SARS-CoV 2 [COVID-19] infection, see Section 10.4.4.1)
    2. Clinically significant pulmonary disease with any 1 pulmonary function parameter < 60% predicted (forced expiratory volume first forced breath [FEV1], total lung capacity [TLC], or diffusing capacity of lungs for carbon monoxide [DLCO]; note: for patients with anemia, corrected DLCO could be used) assessed prior to leukapheresis and within 2 months of the start of lymphodepleting chemotherapy
    3. Requirement for oxygen support (due to cardiac or pulmonary disease)
    4. Interstitial lung disease (pneumonitis) or history of pneumonectomy or chronic obstructive pulmonary disease with ≥ 1 exacerbation within 1 year prior to the Screening Visit that required treatment with systemic corticosteroids or resulted in hospitalization
    5. Hospitalization for bowel obstruction in last 2 months
    6. Hematosis or significant organ bleeding in last 2 months
    7. Ascites or pleural effusion which requires repeated (2 within 4 weeks) paracentesis or thoracentesis within last 2 months
    8. Cardiac or pericardial tumor involvement (prior to lymphodepletion)
11. Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human T cell leukemia virus (HTLV) as defined below. Re-screening for infectious disease markers is not required at baseline (prior to lymphodepletion) unless > 6 months has elapsed.

    1. Positive serology for HIV
    2. Active hepatitis B infection as demonstrated by test for hepatitis B surface antigen. Subjects who are hepatitis B surface antigen negative but are hepatitis B core antibody-positive must have undetectable hepatitis B DNA and receive prophylaxis against viral reactivation. Prophylaxis should be initiated prior to lymphodepleting therapy and continued for 6 months.
    3. Active hepatitis C infection as demonstrated by hepatitis C ribonucleic acid (RNA) test. Subjects who are HCV antibody-positive will be screened for HCV RNA by any reverse transcription-polymerase chain reaction (RT PCR) or branched DNA (bDNA) assay. If HCV antibody is positive, eligibility will be determined based on a negative screening RNA value.
    4. Positive serology for HTLV 1 or 2
12. Subject is pregnant or breastfeeding.
13. Subjects who have illicit drug or alcohol dependency within the past year.
14. In the opinion of the Investigator, subject will be unlikely to fully comply with protocol requirements.
15. Intolerance to nivolumab includes severe allergic reaction to nivolumab or any components (active or inactive) of nivolumab.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the anti-tumor activity of genetically modified autologous T-cells (ADP-A2M4CD8) as monotherapy and in combination with nivolumab in HLA-A*02 positive subjects with MAGE-A4 positive recurrent ovarian cancer | 3.6 years
  Overall Response (OR) is defined as incidence of (confirmed) complete responses or partial responses as assessed by RECIST v1.1 by IRAC from T-cell infusion until documented disease progression

SECONDARY OUTCOMES:
To evaluate safety and tolerability of ADP-A2M4CD8 as monotherapy or in combination with nivolumab | 3.6 years
  Determination of incidence of adverse events and incidence, severity, and duration of AESIs
To evaluate safety of ADP-A2M4CD8 as monotherapy or in combination with nivolumab. | 15 years
  Incidence of patients with Replication-competent Retrovirus, persistence of ADP-A2M4CD8 T-cells and incidence of insertional oncogenesis.
Durable Response (DR) | 3.6 years
  DR per RECIST v1.1 by IRAC and Investigator radiological assessment, defined as a confirmed OR (CR or PR) lasting continuously for 6 months and starting any time within 12 months of T-cell infusion
Time to response (TTR) | 3.6 years
  TTR per RECIST v1.1 by IRAC and Investigator radiological assessment, defined as the duration between the date of T-cell infusion and the initial date of the confirmed response.
Duration of Response (DOR) | 3.6 years
  DoR per RECIST v1.1 by IRAC and Investigator radiological assessment, defined as the duration from the initial date of the confirmed response to the earliest date of PD or death due to any cause.
Progression Free Survival (PFS) | 3.6 years
  PFS per RECIST v1.1 by IRAC and Investigator radiological assessment, defined as the interval between the date of T-cell infusion and the earliest date of disease progression or death due to any cause.
Overall Response (OR) | 3.6 years
  OR is defined as incidence of (confirmed) complete responses or partial responses as assessed by RECIST v1.1 by Investigator radiological assessment from T-cell infusion until documented disease progression
Overall Survival (OS) | 15 years
  OS, defined as the duration between the date of T-cell infusion and the date of death due to any cause.
Levels of serum CA125 | 3.6 years
  Levels of serum CA125 (u/ml) for all patients
Levels of serum CA125 | 3.6 years
  Changes of serum CA125 (u/ml) from baseline for all patients
To characterize the surrogates of treatment effect | 3.6 years
  Peak expansion (DNA copies/μg) (i.e., maximum persistence) by responder status and overall (all patients)
To characterize the surrogates of treatment effect | 3.6 years
  Time to peak expansion (in days since T-cell infusion) by responder status and overall (all patients)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (9):
  - Honor Health, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Augusta University, Augusta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Swedish Cancer Institute, Seattle, Washington
- University Health Network (Princess Margaret Cancer Center), Toronto, Ontario, Canada
- France (4):
  - Institut de Cancerologie des Hospices Civils de Lyon, Pierre-Bénite, Lyon
  - Centre Leon-Berard, Lyon
  - Institut de Cancerologie de Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Spain (7):
  - Vall d'Hebron Unversity Hospital, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Oncologico Clara Campal, Madrid
  - Hospotal Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - University College of London Hospital, London
  - The Christie Hospital, Manchester